CLINICAL TRIAL: NCT05956288
Title: The Hypoalgesic Effects of BFR Training in Nonspecific Shoulder Pain. A Study Protocol of a Crossover Randomized Controlled Clinical Trial
Brief Title: The Hypoalgesic Effects of BFR Training in Nonspecific Shoulder Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Kyriakos Pavlou, PhD student, European University Cyprus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EUC
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Pain; BFR; Shoulder Impingement
Keywords: Shoulder pain; BFR
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood flow restriction (BFR) with low load resistance training (Experimental): A single BFR exercise (Biceps curl with dumbell) will be perform. The initial resistance load for performing the above exercise will correspond to 5% of the body weight of each participant (±0.250 kg). Participants will be asked to perform 4 sets of bicep curls. The first set will consist of repetitions until failure (inability to follow the rhythm or inability to perform an additional contraction) followed by 3 sets of 15 repetitions with 30 seconds rest between sets. In case that for any of the participants will not be able to complete all the repetitions, or they are unable to follow the pace of the metronome, the resistance load will be reduced by 0.5 kg. Vascular Occlusion Pressure will be set at 50-60% of the complete occlusion pressure for the intervention group .Five minutes after the execution of the biceps curl exercise, each participant will receive a specific training which will consist of six therapeutic exercises targeting in loading the rotator cuff and scapula muscles
  Interventions: Device: Blood flow restriction (BFR) with low load resistance training
- Sham-Blood flow restriction (sham-BFR) with low load resistance training (Placebo Comparator): Same procedure as experimental . The only difference between the two groups regarding the intervention will be the percentage of blood flow restriction cuff pressure. In the sham BFR group, as much pressure as 2 fingers can penetrate the cuff will be automatically applied via MADUP®, where based on the literature seems not to promote adaptations related to the use of the method.
  Interventions: Device: Blood flow restriction (BFR) with low load resistance training

INTERVENTIONS:
Device: Blood flow restriction (BFR) with low load resistance training — Combination of low load resistance exercise in the upper limb with the addition of blood flow restriction or sham-blood flow restriction.

SUMMARY:
The primary objective of the present study is to evaluate if a single acute BFR low load- exercise bout would reduce pain in patients with nonspecific shoulder pain and whether the potential hypoalgesia will be maintained after a 45-minute physical therapy shoulder exercise session. BFR exercise will be compared to a sham BFR exercise protocol. We hypothesize that the participants in the BFR group in will experience reduced pain and will be able to complete a scapula and rotator cuff muscles exercise loading program with reduced pain until the end of the exercise program.

DETAILED DESCRIPTION:
Shoulder pathologies are the 3rd most common musculoskeletal condition encountered by health professionals in their day-to-day clinical practice, followed by low back pain and neck pain. It is noteworthy that approximately 40%-54% of patients report ongoing pain lasting between 1-3 years , causing a huge economic burden both on the national health care system but also to the patients. The pathologies associated with development of shoulder pain are numerous, however, in recent years the research community dealing with musculoskeletal shoulder pain has emphasized the need to break free from diagnostic terminologies that refer to precise clinical diagnosis, since such a thig is nearly impossible to happen, due to the low validity and diagnostic accuracy of the special tests available to the clinician. In addition, the need to detach from diagnostic labels becomes even more intense if one takes into account the inability to correlate symptoms and clinical status with pathological findings in diagnostic tests. Nonspecific shoulder pain is an umbrella term that includes non-traumatic musculoskeletal disorders of the shoulder.

Therapeutic exercise is the mainstay of conservative treatment and appears to be a powerful tool in the hands of clinicians to improve pain, mobility, and function of the shoulder in individuals with nonspecific shoulder pain . There are several mechanisms that are hypothesized to explain the benefits of exercise in nonspecific shoulder pain. The neuromuscular mechanism is the most frequently mentioned and is commonly explained as strengthening of the rotator cuff inhibiting pain. Other mechanisms proposed are: tissue factors (e.g. tendon remodeling, blood flow improvement etc.), neuro-endocrine-immune (e.g. exercise induced hypoalgesia, central and peripheral nervous system adaptations etc) and physiological mechanisms (e.g. improvements in self-efficacy and coping with pain etc).

The BFR method is a type of training with parallel partial restriction of arterial inflow and complete venous outflow restriction in muscle tissue that is usually combined with parallel execution of low-load resistance exercises. Blood flow restriction is achieved by using special cuffs applied to both the upper and lower extremities. During the last decade the popularity of this technique seems to be growing rapidly due to its beneficial effects on increasing muscle strength and muscle hypertrophy in healthy adults and clinical population but also its acute hypoalgetic effect on healthy population by significantly increasing the patient pain thresholds. However, to date there is only one published study examining the acute hypoalgetic effects of BFR training in a clinical population, showing beneficial adaptations in reducing pain in people with patellofemoral pain

The primary objective of the present study is to evaluate if a single acute BFR low load- exercise bout would reduce pain in patients with nonspecific shoulder pain and whether the potential hypoalgesia will be maintained after a 45-minute physical therapy shoulder exercise session. BFR exercise will be compared to a sham BFR exercise protocol. We hypothesize that the participants in the BFR group in will experience reduced pain and will be able to complete a scapula and rotator cuff muscles exercise loading program with reduced pain until the end of the exercise program.

ELIGIBILITY:
Adults presenting with nonspecific shoulder pain will be recruited using the following eligibility criteria:

Inclusion Criteria:

* Age >18≤40 years considering that the prevalence for degenerative rotator cuff tendinopathy increases from the age of 40 and above
* Shoulder pain intensity > 4/10 NPRS when performing active glenohumeral abduction and/or isometric resistance to glenohumeral external rotation from 0° of abduction.
* Duration of symptoms > 3 weeks (to avoid an inflammatory clinical picture).

Exclusion Criteria:

* Positive drop arm test (important indication for rotator cuff tear)
* Cervical radiculopathy having a positive specific spurling test or neurological symptoms in the upper limb
* Passive deficit in range of motion (ROM) > 2 levels of motion, where according to the literature it is an indication of frozen shoulder
* Body Mass Index (BMI) > 28
* Previous shoulder surgery
* Previous humerus fracture
* Cancer
* Rheumatic diseases
* Systemic pathologies (e.g. diabetes, rheumatism, fibromyalgia)
* History of previous neurological diseases
* History of thrombosis
* Cardiovascular pathologies
* Neurological diseases
* Long-term use of corticosteroids
* Injury or surgery < 1 month related to the shoulder girdle
* Hypertension (> 140/90mmHg)
* Anti-inflammatory treatment in the last 2 weeks
* Injectable therapy (last 3 months)
* Previous experience/knowledge of the BFR technique
* Inability to write and read Greek

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
Pressure pain detection threshold assessment | Baseline
  PPDT's will assess using a hand-held mechanical pressure algometer in local and remote areas
Pressure pain detection threshold assessment | 15 minutes (1st session)
  PPDT's will assess using a hand-held mechanical pressure algometer in local and remote areas
Pressure pain detection threshold assessment | 1 hour (1st session)
  PPDT's will assess using a hand-held mechanical pressure algometer in local and remote areas
Pressure pain detection threshold assessment | 2nd session (> 72 hours after 1st session)
  PPDT's will assess using a hand-held mechanical pressure algometer in local and remote areas
Pressure pain detection threshold assessment | 15 minutes (2nd session)
  PPDT's will assess using a hand-held mechanical pressure algometer in local and remote areas
Pressure pain detection threshold assessment | 1 hour (2nd session)
  PPDT's will assess using a hand-held mechanical pressure algometer in local and remote areas
Maximal pain and strength in isometric shoulder external rotation | Baseline
  The MVIC of shoulder external rotation will be assessed using a hand held dynamometer. Additionally, the maximum value from 3 successful trials (no >15% difference between the 3 trials) will be used for statistical analysis. In addition, participants will be asked to rate their pain based on the NPRS scale (0-10) during the test.
Maximal pain and strength in isometric shoulder external rotation | 15 minutes (1st session)
  The MVIC of shoulder external rotation will be assessed using a hand held dynamometer. Additionally, the maximum value from 3 successful trials (no >15% difference between the 3 trials) will be used for statistical analysis. In addition, participants will be asked to rate their pain based on the NPRS scale (0-10) during the test.
Maximal pain and strength in isometric shoulder external rotation | 1 hour (1st session)
  The MVIC of shoulder external rotation will be assessed using a hand held dynamometer. Additionally, the maximum value from 3 successful trials (no >15% difference between the 3 trials) will be used for statistical analysis. In addition, participants will be asked to rate their pain based on the NPRS scale (0-10) during the test.
Maximal pain and strength in isometric shoulder external rotation | 2nd session (> 72 hours after 1st session)
  The MVIC of shoulder external rotation will be assessed using a hand held dynamometer. Additionally, the maximum value from 3 successful trials (no >15% difference between the 3 trials) will be used for statistical analysis. In addition, participants will be asked to rate their pain based on the NPRS scale (0-10) during the test.
Maximal pain and strength in isometric shoulder external rotation | 15 minutes (2nd session)
  The MVIC of shoulder external rotation will be assessed using a hand held dynamometer. Additionally, the maximum value from 3 successful trials (no >15% difference between the 3 trials) will be used for statistical analysis. In addition, participants will be asked to rate their pain based on the NPRS scale (0-10) during the test.
Maximal pain and strength in isometric shoulder external rotation | 1 hour (2nd session)
  The MVIC of shoulder external rotation will be assessed using a hand held dynamometer. Additionally, the maximum value from 3 successful trials (no >15% difference between the 3 trials) will be used for statistical analysis. In addition, participants will be asked to rate their pain based on the NPRS scale (0-10) during the test.

SECONDARY OUTCOMES:
Pain during active shoulder Abduction | Baseline (1st session)
  Pain during active shoulder abduction (0 to 180°) in standing in a NPRS scale
Pain during active shoulder Abduction | 15 minutes (1st session)
  Pain during active shoulder abduction (0 to 180°) in standing in a NPRS scale
Pain during active shoulder Abduction | 1 hour (1st session)
  Pain during active shoulder abduction (0 to 180°) in standing in a NPRS scale
Pain during active shoulder Abduction | 2nd session (> 72 hours after 1st session)
  Pain during active shoulder abduction (0 to 180°) in standing in a NPRS scale
Pain during active shoulder Abduction | 15 minutes (2nd session)
  Pain during active shoulder abduction (0 to 180°) in standing in a NPRS scale
Pain during active shoulder Abduction | 1 hour (2nd session)
  Pain during active shoulder abduction (0 to 180°) in standing in a NPRS scale
Patient-perceived pain change | 15 minutes (1st session)
  patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (Jaeschke, 1986)
Patient-perceived pain change | 1 hour (1st session)
  patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (Jaeschke, 1986)
Patient-perceived pain change | 2nd session (> 72 hours after 1st session)
  patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (Jaeschke, 1986)
Patient-perceived pain change | 15 minutes (2nd session)
  patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (Jaeschke, 1986)
Patient-perceived pain change | 1 hour (2nd session)
  patient-perceived pain change using a global rating of change scale (GROC) based on a 7-point Likert scale ranging from "Much better - a very important improvement" to "Much worse - an important aggravation" (Jaeschke, 1986)
Shoulder Pain and Disability Index (SPADI) questionnaire | Baseline
  Shoulder Pain and Disability Index (SPADI) questionnaire which assesses the pain and difficulty experienced by the participant in daily activities of the upper extremity. The questionnaire is translated into Greek and cross-culturally weighted to the Greek population (Vrouva et al., 2016).
Shoulder Pain and Disability Index (SPADI) questionnaire | 2nd session (> 72 hours after 1st session)
  Shoulder Pain and Disability Index (SPADI) questionnaire which assesses the pain and difficulty experienced by the participant in daily activities of the upper extremity. The questionnaire is translated into Greek and cross-culturally weighted to the Greek population (Vrouva et al., 2016).
Participant's rating of perceived exertion (RPE) | 15 minutes (1st session)
  RPE using a modified Borg's scale (Borg CR10) immediately following the blood flow restriction or sham- blood flow restriction exercise session. The scale has been shown to be an valid alternate tool for estimating the exertion and intensity levels during resistance training (Brandt, 2013 ).
Participant's rating of perceived exertion (RPE) | 15 minutes (2nd session)
  RPE using a modified Borg's scale (Borg CR10) immediately following the blood flow restriction or sham- blood flow restriction exercise session. The scale has been shown to be an valid alternate tool for estimating the exertion and intensity levels during resistance training (Brandt, 2013 ).

CONTACTS AND LOCATIONS:
Locations (1):
- European University, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pavlou K, Savva C, Korakakis V, Pamboris GM, Karagiannis C, Ploutarchou G, Constantinou A. Blood Flow Restriction Training in Nonspecific Shoulder Pain: Study Protocol of a Crossover Randomised Controlled Trial. Sports (Basel). 2023 Oct 9;11(10):197. doi: 10.3390/sports11100197. PMID 37888524